CLINICAL TRIAL: NCT02349009
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Topical C-82 in Systemic Sclerosis - A Phase I/II Biomarker and Safety Trial
Brief Title: Trial of Topical C-82 in Systemic Sclerosis - A Phase I/II Biomarker and Safety Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prism Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRI-C82T-3101
Record Dates: First submitted 2015-01-18; First posted 2015-01-28 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2016-09

CONDITIONS: Systemic Scleroderma
Keywords: systemic sclerosis; scleroderma
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): C-82 Topical Gel, Placebo
  Interventions: Drug: C-82 Topical Gel, Placebo
- Active (Active Comparator): C-82 Topical Gel, 1%
  Interventions: Drug: C-82 Topical Gel, 1%

INTERVENTIONS:
Drug: C-82 Topical Gel, 1% — active
  Arms: Active
Drug: C-82 Topical Gel, Placebo — placebo
  Arms: placebo

SUMMARY:
1:1 active treatment: placebo, blinded trial, evaluating the effect of a 4-week treatment period with topical C-82 on skin expression of two gene biomarker surrogates (THBS1 and COMP) for the modified Rodnan skin score (MRSS). Study subjects will be randomized to apply the active study medication daily for 4 weeks to either the right or left forearm and placebo to the contralateral forearm.

DETAILED DESCRIPTION:
1:1 active treatment: placebo, blinded trial, evaluating the effect of a 4-week treatment period with topical C-82 on skin expression of two gene biomarker surrogates (THBS1 and COMP) for the modified Rodnan skin score (MRSS). Study subjects will be randomized to apply the study medication daily for 4 weeks to either the right or left forearm. All subjects will apply placebo (i.e., a topical gel without C-82) to the contralateral forearm. Both physician and subject will be blinded to treatment arm assignment. Skin biopsies will be taken from the mid-forearm of both arms at baseline and after four weeks of study drug to test for biomarker gene expression; instructions and supplies will be provided to each site. Safety assessments will extend to 4 weeks after the final dose of study drug/placebo.

ELIGIBILITY:
Inclusion Criteria:

* meet the American College of Rheumatology criteria for systemic sclerosis with diffuse cutaneous involvement (clinical skin involvement proximal to forearms and or knees, not including the face).
* Disease duration of <36 months since the onset of the first SSc manifestation other than Raynaud's phenomenon, or patients with progressive disease based on new or worsening skin disease based on physician assessment.
* local skin score over the bilateral forearm of ≥ 2.
* a MRSS of ≥ 12.
* on stable dose of any immunosuppressive other than cyclophosphamide or high dose steroids (excluded treatments) for at least one month and through the course of study treatment.
* Subjects of child-producing potential must agree to use effective contraception while and for at least 3 months after the last treatment.

Exclusion Criteria:

* Receiving treatment as part of an interventional clinical trial within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer).
* Ongoing use of high dose steroids (> 10mg/day prednisone or equivalent) or unstable steroid dose in the past 4 weeks.
* Use of topical creams or gels on the forearm area within the past month and through the course of study treatment.
* UV light therapy for 4 weeks before or during the study period.
* Treatment with cyclophosphamide within the past month and through the course of study treatment.
* Known active bacterial, viral fungal mycobacterial, or other infection
* history of malignancy within the past 2 years.
* Moderate to severe hepatic impairment, .
* Scleroderma renal crisis within 4 months or creatinine greater than 2.0.
* Pregnancy.
* Nursing mothers are to be excluded.
* Gastrointestinal involvement requiring total parenteral nutrition or hospitalization within the past 3 months for pseudo-obstruction
* Moderately severe pulmonary disease with FVC < 40%, or DLCO < 30% predicted or evidence of progressive lung disease as manifest by a decrease in FVC or 10% or more over the previous year.
* Moderately severe cardiac disease with clinically significant heart failure, or unstable angina.
* AST or ALT > 2.5 x Upper Limit of Normal.
* Total bilirubin > 1.5 x upper limit of normal (ULN). Patients with Gilbert's Disease may be included if their total bilirubin is ≤ 3.0 mg/dL.
* significant medical or psychosocial problems that warrant exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
frequency and character of adverse events and abnormal clinical tests | 28 days
change in gene biomarker expression of THBS1 and COMP in skin biopsies over time compared to placebo | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lafyatis, MD, Principal Investigator — Boston University
Locations (3):
- United States (3):
  - Chicago, Illinois
  - Boston, Massachusetts
  - New York, New York